CLINICAL TRIAL: NCT04731272
Title: Effect of GLP-1 Agonist Therapy on Insulin Secretion in Adults With Pancreatic Insufficient Cystic Fibrosis and Abnormal Glucose Tolerance: a Randomized, Open-label, Cross-over Trial
Brief Title: GLP-1 Agonist Therapy in Cystic Fibrosis-Related Glucose Intolerance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Michael R. Rickels, MD, MS, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 848357
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency; Abnormal Glucose Tolerance; Diabetes
Keywords: Cystic Fibrosis Related Diabetes; Glucose Intolerance; Insulin Secretion; Glucagon-Like Peptide-1 (GLP-1)
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Diabetes Mellitus; Glucose Intolerance | interventions — dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dulaglutide (Experimental): The Mixed Meal Tolerance Test as described in the primary outcome section will be performed at baseline and after 6 weeks of dulaglutide therapy in the intervention period.
  Interventions: Drug: Dulaglutide 0.75Mg/0.5Ml Inj Pen
- Observation (No Intervention): The Mixed Meal Tolerance Test as described in the primary outcome section will be performed at baseline and after 6 weeks of no intervention in the observation period.

INTERVENTIONS:
Drug: Dulaglutide 0.75Mg/0.5Ml Inj Pen — Randomized, open-label, cross-over study of 6 weeks exposure to dulaglutide 0.75 mg subcutaneous weekly or observation.
  Arms: Dulaglutide

SUMMARY:
Diabetes is a major co-morbidity in pancreatic insufficient cystic fibrosis (PI-CF) and associated with worse outcomes. While reduced β-cell mass contributes to the insulin secretory defects that characterizes cystic fibrosis-related diabetes (CFRD), other modifiable determinants appear operative in the emergence and progression of abnormal glucose tolerance towards diabetes. Identifying interventions to preserve β-cell function are crucial for delaying and potentially preventing CFRD development. In this study, we hypothesize that weekly administration of the long-acting glucagon-like peptide-1 (GLP-1) agonist dulaglutide will improve defective early-phase insulin secretion and improve glucose tolerance during a mixed-meal tolerance test.

DETAILED DESCRIPTION:
Diabetes is a major co-morbidity in pancreatic insufficient cystic fibrosis (PI-CF) and associated with worse outcomes. While reduced β-cell mass contributes to the insulin secretory defects that characterizes cystic fibrosis-related diabetes (CFRD), other modifiable determinants appear operative in the emergence and progression of abnormal glucose tolerance towards diabetes. Identifying interventions to preserve β-cell function are crucial for delaying and potentially preventing CFRD development. In this study, we hypothesize that weekly administration of the long-acting glucagon-like peptide-1 (GLP-1) agonist dulaglutide will improve defective early-phase insulin secretion and improve glucose tolerance during a mixed-meal tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, aged ≥18 years on date of consent
* 2. Confirmed diagnosis of CF, defined by positive sweat test or Cystic Fibrosis transmembrane conductance regulator (CFTR) mutation analysis according to Cystic Fibrosis Foundation (CFF) diagnostic criteria.
* 3. Pancreatic insufficiency defined by clinical requirement for pancreatic enzyme replacement.
* 4. Abnormal glucose tolerance defined by OGTT criteria for EGI, IGT, or CFRD, or diagnosed CFRD.

  1. There will be no restriction on enrollment of individuals with CFRD but without fasting hyperglycemia (fasting hyperglycemia is defined as fasting glucose ≥126 mg/dL)
  2. Individuals with CFRD and fasting hyperglycemia (defined as above or by the use of basal insulin therapy) must also have a HbA1c ≤8% and a random (non-fasting) C-peptide ≥1.2 ng/mL17; enrollment of this subgroup will be limited to n =10.
* 5. Ability to take subcutaneous medication and be willing to adhere to the weekly administration regimen and complete study specific procedures (MMTT)
* 6. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 6 weeks after the end of dulaglutide or observation administration; oral contraceptives, intra-uterine devices, Norplant®, Depo-Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable

Exclusion Criteria:

* 1. BMI <19 kg/m2
* 2. Presence of first-degree atrioventricular block or other evidence for cardiac conduction system or structural heart defects
* 3. Pregnancy or lactation; a negative urine pregnancy test will be required at enrollment
* 4. Known allergic reactions to any GLP-1 agonist, and any history of severe hypersensitivity reactions (anaphylaxis or angioedema)
* 5. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome type 2 (MEN2)
* 6. Pulmonary exacerbation requiring IV antibiotics or systemic glucocorticoids within 4 weeks prior to study procedures
* 7. Gastrointestinal symptom exacerbation defined by current nausea/vomiting or diarrhea
* 8. Established diagnosis of non-CF diabetes (e.g. type 1 diabetes) or CFRD with fasting hyperglycemia (fasting glucose ≥126 mg/dL [use of prandial insulin or repaglinide will be permitted])
* 9. History of clinically symptomatic pancreatitis within the last year
* 10. Prior lung, liver or other solid organ transplant
* 11. Severe CF liver disease, as defined by the presence of portal hypertension
* 12. History of fundoplication-related dumping syndrome
* 13. Hemoglobin <10 g/dL, within 90 days of study procedures or at screening
* 14. Abnormal renal function, within 90 days of study procedures or at screening; defined as creatinine >2x upper limit of normal (ULN) or potassium >5.5mEq/L on non-hemolyzed specimen
* 15. History of any illness or condition that, in the opinion of the investigator might confound the results of the study or pose an additional risk to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Early-phase insulin secretion | 18 weeks
  The primary outcome measure is the insulin secretory rate during the first 30-min during a mixed meal tolerance test (ISR-AUC30).

SECONDARY OUTCOMES:
Early-phase insulin secretion adjusted for glucose excursion | 18 weeks
  This secondary outcome measure is insulin secretory rate/glucose area under cure during the first 30-min during a mixed meal tolerance test (ISR-AUC30/ Glc-AUC30)
Glucose tolerance | 18 weeks
  This secondary outcome measure is mixed meal tolerance test-related glucose area under the curve over 180 min (Glc-AUC180).

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Rickels, MD, MS, Principal Investigator — University of Pennsylvania; Andrea Kelly, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Colorado, Aurora, Colorado
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of enrollment.
Supporting Information: ICF
Time Frame: Upon completion of enrollment.
Access Criteria: Consent will be uploaded to CT.gov